CLINICAL TRIAL: NCT07345078
Title: Study on the Treatment of Post-stroke Dysphagia and Stroke-associated Pneumonia With Bronchoscopy
Acronym: Sottopdaspwb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Zunyi (Other)
Responsible Party: Principal Investigator, Huajun Yang, Associate Chief Physician, The First People's Hospital of Zunyi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZ（2019）146
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Stroke Associated Pneumonia; Non Severe Ischemic Stroke; Dysphagia
Keywords: bronchoscope
MeSH Terms: conditions — Deglutition Disorders | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Intervention Model Description: The control group was given conventional anti-infective drugs, expectorants, and suctioning with a suction tube. The treatment group was treated with fiberoptic bronchoscopy for sputum suction and bronchoalveolar lavage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received routine anti-infection and expectorant treatment and was given suctioning with a suction tube as needed, that is, suctioning at any time when breathing is difficult or there is a sound of phlegm in the airway.
- Observation group (Experimental): The observation group received 1-2 sessions of bronchoscopy treatment, including suction, lavage, and medication injection under the microscope. Two groups were treated continuously for one week.
  Interventions: Device: Tracheoscopy suction and bronchoalveolar lavage

INTERVENTIONS:
Device: Tracheoscopy suction and bronchoalveolar lavage — On the basis of the control group, the observation group received 1-2 sessions of bronchoscopy treatment, including suction, lavage, and medication injection under the microscope. Specific operating steps: Use atropine injection 0.5 mg combined with lidocaine injection 0.1 g nebulized inhalation for local anesthesia. The Olympus BF-P180 fiberoptic bronchoscope is routinely inserted through the nasal cavity and sequentially enters each level of bronchus to clean airway secretions under direct vision. Collect lavage fluid for bacterial culture and drug sensitivity testing. When the sputum is thick and difficult to aspirate, physiological saline can be used for lavage. Both groups are treated continuously for one week.
  Other Names: Tracheoscopy suction; bronchoalveolar lavage
  Arms: Observation group

SUMMARY:
Select 50 non-severe ischemic SAP patients with swallowing difficulties in our intensive care unit and randomly divide them into two group.The control group was given conventional anti-infective drugs, expectorants, and suctioning with a suction tube. The treatment group was treated with fiberoptic bronchoscopy suction and bronchoalveolar lavage, while the drug treatment was the same as the control group. Compare heart rate, respiration, blood pressure, blood oxygen saturation, arterial blood gas analysis, procalcitonin, interleukin-32, lung function, C-reactive protein, clinical pulmonary infection score (CPIS), swallowing difficulty assessment scale, and adverse reactions between two groups.

DETAILED DESCRIPTION:
Stroke-associated pneumonia (SAP) is one of the most common respiratory complications of acute stroke, which occurs in about 4% to 9% of patients after stroke. Among patients with acute ischemic stroke who receive treatment in the neurological intensive care unit and those who need feeding through a nasogastric tube, the incidence rate of stroke-associated pneumonia is higher (21% and 44%, respectively). Compared with patients without pneumonia, stroke-related pneumonia patients have a higher mortality rate and poorer long-term prognosis. Pneumonia is the most common cause of fever within 48 hours after acute stroke and also the most common complication within 2-4 weeks after supratentorial ischemic infarction. In addition, retrospective data indicate that pneumonia and respiratory diseases are the most common causes of hospitalization among stroke survivors in the first five years after ischemic stroke. The independent risk factors for hospitalized pneumonia are age over 65 years, articulation disorders or speechlessness caused by aphasia, severe post-stroke disability, cognitive impairment, and swallowing difficulties. In an early prospective study, the risk factors for 124 acute stroke patients receiving treatment in the intensive care unit were mechanical ventilation, abnormal chest X-rays upon admission, and swallowing difficulties. Post-stroke aspiration pneumonia is usually caused by stroke-related swallowing difficulties (i.e., impaired swallowing motor and sensory mechanisms) or decreased consciousness leading to impaired cough reflex and glottal closure. Moreover, prophylactic use of antibiotics in acute stroke patients cannot reduce the incidence of post-stroke pneumonia or improve prognosis.

Dysphagia is a common symptom of end-stage illness, where a decline in swallowing function during the last weeks to months of life weakens people's desire and ability to eat. Dysphagia of solids and liquids is one of the most common symptoms in the last few days of life. Dysphagia can affect quality of life (such as socializing and communication), leading to nutritional and water intake disorders. Dysphagia is also a major susceptible inhalation condition and can cause pneumonia, and in some cases, even suffocation or death. Considering that food and nutrition are the central focus of social interaction, as well as people's general concern for the nutrition needed for health, swallowing disorders can also bring setbacks and pain to home caregivers and healthcare workers. In addition, for many end-stage disease patients, inability to swallow and/or disinterest in food may be a key symptom that prompts them to decide to give up treatment and end-of-life care. Dysphagia refers to difficulty swallowing food or liquids, including medications in liquid or pill form. Dysphagia after stroke may be caused by motor or sensory dysfunction in neural processes, which can lead to problems with eating certain types of food or liquids, or even inability to swallow at all. Patients may complain about food getting stuck in the upper digestive tract from the throat to the distal esophagus and experiencing coughing or suffocation while eating or drinking. Chronic swallowing difficulties can affect the efficiency of oral feeding, leading to physical weakness, decreased appetite, weight loss, dehydration, and malnutrition. In addition, airway protection or swallowing safety may also be threatened by swallowing disorders. Food or liquids may transfer into the trachea, causing inhalation, suffocation, or, in severe cases, suffocation. Inhalation Pneumonia is an infectious process caused by inhalation of oral and pharyngeal secretions colonized by pathogenic bacteria. Gram-negative Escherichia coli and anaerobic bacteria are the most common pathogenic microorganisms, while inhalation of sterile acidic gastric contents can also cause acute chemical damage to the lungs. Therefore, improving dysphagia after stroke is particularly important for the treatment of SAP, which can remove the etiology, significantly reduce the incidence rate of SAP, and improve the prognosis. Swallowing is not a random activity but a complex reflex activity that requires specific stimuli to trigger. Although swallowing can be initiated at will, the process of completing this action is a complex reflex activity. A simple swallowing movement requires coordination of 25 pairs of muscles in the mouth, pharynx, larynx, esophagus, and face, with the participation of at least 6 pairs of cranial nerves, language, and respiratory systems. Swallowing is a typical and complex reflex action that involves a series of sequential steps, each consisting of a series of activity processes, where the activity of the previous step can trigger the activity of the subsequent step. The receptors for swallowing activity are located in the soft palate, posterior pharyngeal wall, epiglottis, and esophagus. Their afferent nerves include fibers from the soft palate (5th and 9th pairs), posterior pharyngeal wall (9th pair), epiglottis (10th pair), and esophagus (10th pair of cranial nerves). The basic center is located in the medulla oblongata, and the efferent nerves are located in the 5th, 9th, 10th, 11th, and 12th pairs of cranial nerves. Their effector organs include muscle groups such as the tongue, throat, pharyngeal muscles, and esophagus. Every step of swallowing is interconnected and indispensable. After a stroke, if the lesion affects the medulla oblongata, swallowing and breathing difficulties may occur.

Domestic research mainly focuses on prevention of SAP-related risk factors, cluster nursing, rehabilitation training, and acupuncture and moxibustion treatment of traditional Chinese medicine, but there is no report on the treatment of dysphagia after stroke by tracheoscopy. Bedside bronchoscopy can clear airway secretions directly through the glottis, stimulate coughing and swallowing muscles to produce contraction movements, and play a positive role in preventing aspiration and relieving swallowing difficulties. Tracheoscopy can directly stimulate the trigeminal nerve of the soft palate, the glossopharyngeal nerve of the posterior pharyngeal wall, and the vagus nerve of the epiglottis, promoting the contraction movement of the chewing muscle group, suprahyoid muscle group, infrahyoid muscle group, facial muscle, tongue muscle, and soft palate muscle group, thereby training the swallowing muscle group, exercising swallowing function, improving swallowing disorders, and significantly reducing the incidence and mortality of SAP.

At present, there are no reports of bedside bronchoscopy for the treatment of post-stroke dysphagia and SAP at home and abroad. This study attempts to explore the application value and clinical safety of portable fiberoptic bronchoscopy (bronchoscope) in non-severe SAP dysphagia patients and evaluate whether bronchoscopy treatment can alleviate the symptoms of dysphagia in SAP patients and improve hypoxia, pulmonary infection, and SAP prognosis.

After obtaining the consent of the subjects, 50 non-severe ischemic SAP patients with swallowing difficulties in our intensive care unit were selected and randomly divided into a treatment group and a control group using a random number table method. The control group was given conventional anti-infective drugs, expectorants, and suctioning with a suction tube. The treatment group was treated with fiberoptic bronchoscopy suction and bronchoalveolar lavage, while the drug treatment was the same as the control group. Compare heart rate, respiration, blood pressure, blood oxygen saturation, arterial blood gas analysis, procalcitonin, interleukin-32, lung function, C-reactive protein, clinical pulmonary infection score (CPIS), swallowing difficulty assessment scale, and adverse reactions between two groups. Comparing the advantages of bronchoscopic sputum aspiration and bronchoalveolar lavage treatment for subjects, direct stimulation of the glottis and pharynx through bronchoscopy induces afferent impulses in neurons (V, VII, X, XII), triggering coughing and Pharyngeal muscle contraction enables pharyngeal muscle exercise, improves swallowing difficulties, reduces aspiration, gradually restores diet, and enhances body function Nurture and promote recovery.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for acute stroke and is clearly diagnosed through head MRI or CT examination.
* According to the Wada drinking water test, there is indeed difficulty swallowing.
* Pneumonia occurs within 72 hours after stroke, confirmed by chest imaging examination, and meets the diagnostic criteria for stroke-related pneumonia.
* Clear consciousness, stable vital signs, and able to cooperate with bronchial examination.

Exclusion Criteria:

* The condition is critical, with severe hemiplegia and mental disorders that cannot tolerate bronchoscopy treatment.
* Combined lung tumors, open pulmonary tuberculosis, coagulation dysfunction, severe cardiovascular and cerebrovascular diseases, severe heart, liver, and kidney dysfunction, and pulmonary infection before stroke.
* Not willing to undergo bronchoscopy examination.
* Individuals with previous esophageal functional structural abnormalities.
* Disagree with participating researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
NIHSS scores | From enrollment to the end of treatment at 2 weeks.
  It is a standardized tool used to assess the degree of neurological deficits in patients with acute stroke, consisting of 15 items covering consciousness level, visual field, facial paralysis, limb movement, ataxia, sensory, language, and articulation disorders. The scoring range for each project is 0 to 4 points, with 0 indicating no defects and higher scores indicating more severe neurological deficits; The total score ranges from 0 to 42 points, with 0 indicating no neurological deficits and 42 indicating extremely severe deficits
Acute Physiology and Chronic Health Evaluation (APACHE) II scores | From enrollment to the end of treatment at 2 weeks.
  It includes three parts: acute physiology score (APS), chronic physiology score (CPS), and patient age score, with a total score of 0-71 points. The higher the score, the more severe the patient's condition, the worse the prognosis, and the higher the mortality rate
CPIS scores | From enrollment to the end of treatment at 2 weeks.
  Clinical Pulmonary Infection Scores
Water Swallow Test scores | From enrollment to the end of treatment at 2 weeks.
  Grade I: able to drink without coughing within 5 seconds; Grade II: No coughing after drinking twice or more; Grade III: Can be consumed in one go but accompanied by coughing; Grade IV: Drink twice or more with coughing; Grade V: Frequent coughing and inability to finish all drinks. Grade I indicates normal, Grade II indicates suspicious, and Grade III or above indicates abnormal.
CRP | From enrollment to the end of treatment at 2 weeks.
  C-reactive protein
Length of hospital stay | From enrollment to the end of treatment at 4 weeks.
  The length of hospital stay from enrollment to discharge
PaO2 | From enrollment to the end of treatment at 2 weeks.
  Arterial partial pressure of oxygen
Height | From enrollment to the end of treatment at 1 week.
  Subject's height（m）
Weight | From enrollment to the end of treatment at 1 week.
  Subject's weight（Kg）
BMI | From enrollment to the end of treatment at 1 week.
  Body Mass Index (Report BMI in kg/m² by combining weight and height)

CONTACTS AND LOCATIONS:
Locations (1):
- Zunyi First People's Hospital, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
ICMJE journals and other team members involved in the research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT07345078/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT07345078/ICF_001.pdf